CLINICAL TRIAL: NCT00957411
Title: Phase II Randomized Assessing Pelvic Irradiation Combined With Cisplatin Alone or Cisplatin Plus Cetuximab in Patients With Carcinoma of the Cervix Stage IB2, II and III
Brief Title: Radiation Therapy and Cisplatin With or Without Cetuximab in Treating Patients With Stage IB, Stage II, or Stage IIIB Cervical Cancer
Acronym: CETUXICOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000651250; CLCC-IC-2007-04 (Other: Institut Curie); 2008-001053-18 (EudraCT Number)
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cervical Cancer
Keywords: stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; cervical adenocarcinoma; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cetuximab; Cisplatin

ARMS (2):
- Arm I (Active Comparator): Patients receive cisplatin IV over 1 hour once weekly during weeks 1-6. Patients also undergo pelvic radiotherapy 5 days a week during weeks 2-5 or 2-6.
  Interventions: Drug: cisplatin
- Arm II (Experimental): Patients receive cisplatin and undergo radiotherapy as in arm I. Patients also receive cetuximab IV over 1 hour once weekly during weeks 1-6.
  Interventions: Biological: cetuximab; Drug: cisplatin

INTERVENTIONS:
Biological: cetuximab — Given IV
  Arms: Arm II
Drug: cisplatin — Given IV

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether radiation therapy given together with cisplatin is more effective with or without cetuximab in treating patients with cervical cancer.

PURPOSE: This randomized phase II trial is studying giving radiation therapy together with cisplatin to see how well it works compared with radiation therapy and cisplatin given together with cetuximab in treating patients with stage IB, stage II, or stage IIIB cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of treatment with cetuximab and a standard radiochemotherapy regimen (pelvic radiotherapy and cisplatin) in patients with stage IB2, II, and IIIB cervical cancer by evaluating the number of patients without recurrence at 2 years.

Secondary

* Analyze the tumor response by MRI after external radiotherapy.
* Assess the tolerance of cetuximab and standard radiochemotherapy in patients not previously treated and in generally good condition.
* Study the correlation between treatment response and analysis of EGFR mutations (exons 18-21 of the tyrosine kinase domain including the two hot spots L858R and E746-A750).
* Study the correlation between treatment response and evaluation of number of copies of the EGFR gene.
* Study the correlation between treatment response and analysis of mutations of codons 12 and 13 of KRAS2 by direct sequencing.
* Study the correlation between treatment response and research of DNA sequences of human papillomavirus.
* Study the correlation between treatment response and overexpression of EGFR and COX2 (centralized) by IHC.
* Study the correlation between treatment response and characterization of a genomic signature (genome, transcriptome, and Affymetrix chips from samples frozen in liquid nitrogen).
* Collect tumor samples for molecular analysis.

OUTLINE: This is a multicenter study. Patients are stratified according to planned surgery (yes vs no) and are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cisplatin IV over 1 hour once weekly during weeks 1-6. Patients also undergo pelvic radiotherapy 5 days a week during weeks 2-5 or 2-6.
* Arm II: Patients receive cisplatin and undergo radiotherapy as in arm I. Patients also receive cetuximab IV over 1 hour once weekly during weeks 1-6.

After 6-8 weeks of study treatment, patients continue treatment as recommended by their center (i.e., utero-vaginal brachytherapy, additional radiotherapy, or surgery).

Tumor tissue and blood samples are collected for further analysis.

After completion of study treatment, patients are followed at 3-4 weeks and then every 4 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cervical cancer

  * Squamous cell carcinoma or adenocarcinoma
  * Stage IB2-IIIB disease
  * Not immediately operable
* Origin of the tumor and presence of measurable target lesion according to RECIST criteria confirmed by T2-weighted MRI
* Data imaging scan and PET scan (optional) confirmed absence of lumbo-aortic adenopathy
* No other associated pathology that would preclude study treatment

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin > 10 g/dL
* ANC > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Alkaline phosphatase < 2 times normal
* Total bilirubin < 1.5 times normal
* Creatinine < 130 μmol/L
* Creatinine clearance ≥ 60 mL/min
* Normal vital functions
* Not pregnant
* Fertile patients must use effective contraception
* Able to provide the imaging exams on CD ROM (DICOM 3.0 or higher) for centralized review
* No history of another cancer that recurred within the past 5 years except for basal cell carcinoma of the skin or carcinoma in situ of the cervix
* No absolute contraindication to MRI (i.e., claustrophobia, pacemaker, or cochlear implant)
* No geographical, social, or psychological situations that preclude study follow up
* Not deprived of liberty or under guardianship
* Receiving benefits from a social security system

PRIOR CONCURRENT THERAPY:

* No prior treatment (i.e., chemotherapy, radiotherapy, immunotherapy, hormonal therapy, or, especially, therapy with an investigational agent) for this cancer
* No concurrent participation in a clinical trial with an experimental agent

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-03; Primary Completion 2013-11 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Recurrence-free survival at 2 years

SECONDARY OUTCOMES:
Response as assessed by MRI after radiochemotherapy and before surgery according to RECIST criteria
Toxicity according to NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Susan Scholl, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie Hopital, Paris, France

REFERENCES:
- [Result] de la Rochefordiere A, Kamal M, Floquet A, Thomas L, Petrow P, Petit T, Pop M, Fabbro M, Kerr C, Joly F, Sevin E, Maillard S, Cure H, Weber B, Brunaud C, Minsat M, Gonzague L, Berton-Rigaud D, Aumont M, Gladieff L, Peignaux K, Bernard V, Leroy Q, Bieche I, Margogne A, Nadan A, Fourchotte V, Diallo A, Asselain B, Plancher C, Armanet S, Beuzeboc P, Scholl SM. PIK3CA Pathway Mutations Predictive of Poor Response Following Standard Radiochemotherapy +/- Cetuximab in Cervical Cancer Patients. Clin Cancer Res. 2015 Jun 1;21(11):2530-7. doi: 10.1158/1078-0432.CCR-14-2368. Epub 2015 Feb 27. PMID 25724520